CLINICAL TRIAL: NCT04649385
Title: A Phase 1 Study Investigating the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of HPK1 Inhibitor BGB-15025 Alone and in Combination With Anti-PD-1 Monoclonal Antibody Tislelizumab in Patients With Advanced Solid Tumors
Brief Title: BGB-15025 Alone and in Combination With Anti-PD-1 Monoclonal Antibody Tislelizumab in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-15025-101; CTR20212721 (Other: ChinaDrugTrials)
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): Part A: Participants will receive once daily of BGB-15025 monotherapy in sequential cohorts of approximately 7 increasing doses
  Part B: Participants will receive once daily of BGB-15025 in sequential cohorts plus 200mg tislelizumab on day 1 of each 21-day cycle (combination therapy )
  Interventions: Drug: BGB-15025; Drug: Tislelizumab
- Phase 1b: Dose Expansion (Experimental): Phase 1b dose expansion will begin based upon the recommended doses for expansion (RDFE) for BGB-15025 alone or in combination with tislelizumab, and with or without chemotherapy as determined from Phase 1a
  Interventions: Drug: BGB-15025; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-15025 — Administered orally once or twice daily (QD or BID)
Drug: Tislelizumab — Administered 200 mg intravenous (IV) infusion
  Other Names: BGB-A317

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of BGB-15025 alone and in combination with tislelizumab; and to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and recommended Phase 2 doses (RP2D) of BGB-15025 alone and in combination with tislelizumab in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Phase 1a (dose escalation): Participants with histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors who have previously received standard systemic therapy or for whom treatment is not available, not tolerated or refused, and who have not received prior therapy targeting HPK1
2. Phase 1b (dose expansion): Participant with histologically or cytologically confirmed advanced, metastatic, and unresectable solid tumors, including non-small cell lung cancer, esophageal cancer or gastric/Gastroesophageal junction cancer (other solid tumors may be included) who have progressed following systemic anticancer therapies or have no prior systemic treatment for advanced disease
3. At least 1 measurable lesion as defined per RECIST 1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
5. Adequate organ function as indicated by the following laboratory values up to first dose of study treatment: Hemoglobin≥ 90 g/L, Absolute neutrophil count ≥ 1.5 x 109/L , Serum total bilirubin ≤ 1.5 x ULN (< 3 x ULN for participants with Gilbert syndrome ), AST and ALT≤ 2.5 x ULN

Key Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled and untreated brain metastasis.
2. Active autoimmune diseases or history of autoimmune diseases that may relapse
3. Any active malignancy ≤ 2 years before the first dose of study treatment except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent
4. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study treatment
5. History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including but not limited to pulmonary fibrosis, acute lung diseases, etc.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of participants with dose limiting toxicities (DLTs) | Up to 3 Years
  Participants will be considered evaluable for DLTs if they 1) received ≥ 80% of each scheduled study treatment administration during the DLT assessment window and/or 2) experienced a DLT.
Phase 1a: Number of Participants Experiencing Adverse Events (AEs) | Up to 4 Years
Phase 1a: Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 4 years
The maximum tolerated dose (MTD) of BGB-15025 | Up to 3 Years
  The highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30%
Recommended Doses for Expansion (RDFE) of BGB-15025 monotherapy | Up to 3 years
  The highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30%
RDFE of BGB-15025 in combination with tislelizumab | Up to 3 years
  The highest dose evaluated for which the estimated toxicity rate is closest to the target toxicity rate of 30%
Phase 1b: Overall Response Rate (ORR) as assessed by the investigator | Up to 2 years

SECONDARY OUTCOMES:
Phase 1a: Overall Response Rate (ORR) as assessed by the investigator | Up to 3 years
Duration Of Response (DOR) as assessed by the investigator | Up to 3 years
Disease Control Rate (DCR) as assessed by the investigator | Up to 3 years
Phase 1a: Maximum observed plasma concentration (Cmax) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Minimum observed plasma concentration (Cmin) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Time to maximum plasma concentration (Tmax) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Half-life of (t1/2) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Area under the concentration-time curve (AUC) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Apparent clearance (CL/F) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Apparent volume of distribution (Vz/F) of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Accumulation Ratio for Cmax of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Accumulation Ratio for AUC of BGB-15025 | Predose up to 8 hours postdose
Phase 1a: Metabolite to parent ratio for BGB-15025 and its metabolite | Predose up to 8 hours postdose
Phase 1b: Number of Participants Experiencing Adverse Events (AEs) | Up to 3 years
Phase 1b: Number of Participants Experiencing Serious Adverse Events (SAEs) | Up to 3 years
Phase 1b: Plasma Concentrations of BGB-15025 | Predose up to 8 hours postdose
Phase 1b: Plasma Concentrations of the metabolite | Predose up to 8 hours postdose
Phase 1b: Number of participants with dose limiting toxicities (DLTs) | Up to 1 year
  Participants will be considered evaluable for DLTs if they 1) received ≥ 80% of each scheduled study treatment administration during the DLT assessment window and/or 2) experienced a DLT.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (3):
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Ut Health San Antonio Mays Cancer Center, San Antonio, Texas
- Australia (4):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Ashford Cancer Centre Research Northeast, Windsor Gardens, South Australia
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (7):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes